CLINICAL TRIAL: NCT01403701
Title: Effects of Physical Therapy on Quality of Life and Function Following Vaginal Reconstructive Surgery; a Randomized Trial
Brief Title: Physical Therapy on Quality of Life and Function Following Vaginal Surgery Reconstructive Surgery
Acronym: PT and QOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09015-09-020
Record Dates: First submitted 2011-07-21; First posted 2011-07-27 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Quality of Life; Pelvic Floor Distress and Impact Scores; Sexual Function Scores
Keywords: physical therapy; pelvic prolapse; incontinence; quality of life
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical therapy (Experimental): Standardized pelvic floor physical therapy
  Interventions: Behavioral: Physical therapy
- routine care (No Intervention): Standard postoperative visits

INTERVENTIONS:
Behavioral: Physical therapy — pelvic floor physical therapy
  Arms: Physical therapy

SUMMARY:
i) The primary objective of this study is to determine if physical therapy improves postoperative quality of life in participants following vaginal reconstructive surgery for pelvic organ prolapse and urinary incontinence.

ii) Secondary objectives include:

1. Comparing pelvic floor symptoms (urinary symptoms, defecatory symptoms and prolapse symptoms) in participants undergoing physical therapy compared to standard postoperative care
2. Comparing sexual function in participants undergoing physical therapy compared to standard postoperative care;
3. Comparing postoperative pain scales, and activity assessment in participants undergoing physical therapy compared to standard postoperative care;
4. Comparing pelvic floor strength and pelvic organ prolapse quantification (POPQ)(12) in participants undergoing physical therapy compared to standard postoperative care.

DETAILED DESCRIPTION:
This is a single center randomized controlled trial assessing quality of life in participants following vaginal surgery receiving physical therapy compared to standard postoperative care. Patients will be under care of the physicians of the Division of Urogynecology and Reconstructive Pelvic Surgery. All physicians are board certified, fellowship trained urogynecologists.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal reconstructive surgery for prolapse
* Age of at least 18 years
* Willing to comply with physical therapy

Exclusion Criteria:

* i. Use of mesh/graft material during the prolapse repair
* ii. Abdominal or laparoscopic prolapse repair
* iii.Current genitourinary fistula or urethral diverticulum
* iv. Contraindication to surgery
* v. Unable to comply with physical therapy or office visits
* vi. Preexisting neurological condition
* vii.Concurrent surgery for fecal incontinence

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-07; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
postoperative quality of life as based on the scores of the WHO-QOL Bref in participants following vaginal reconstructive surgery for pelvic organ prolapse and urinary incontinence | 3-6 months
  Quality of life scores on the world health organization validated quality of life scale

SECONDARY OUTCOMES:
Comparing pelvic floor quality of life scores and distress related to pelvic floor symptoms (urinary symptoms, defecatory symptoms and prolapse symptoms) in participants undergoing physical therapy compared to standard postoperative care | 3-6 months
  several validated indices for measuring symptoms of urinary and bowel symptoms
Comparing sexual function scores in participants undergoing physical therapy compared to standard postoperative care; | 3-6 months
  based on validated indices of sexual function

CONTACTS AND LOCATIONS:
Overall Officials: Rachel N Pauls, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- TriHealth, Inc, Cincinnati, Ohio, United States